CLINICAL TRIAL: NCT06835712
Title: Virtual Reality and Guided Imagery to Reduce Pain During Peripheral Intravenous Catheterization Procedure in Adults: A Randomized Controlled Trial
Brief Title: Virtual Reality and Guided Imagery to Reduce Procedural Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Derya Uzelli, Associate Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0040
Record Dates: First submitted 2025-02-08; First posted 2025-02-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pain Management; Virtual Reality Pain Distraction; Guided Imagery; Peripheral Intravenous Catheterization Application
Keywords: virtual reality; guided imagery; pain management; peripheral intravenous catheterization
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The virtual reality group (Experimental): During peripheral intravenous catheterization, virtual reality headset (Oculus Go) will be worn. Because the headset is reusable, attention will be paid to disinfecting them before and after each use.
  Interventions: Other: The guided imagery
- The guided imagery group (Experimental): During peripheral intravenous catheterization, an audio clip Mp3 player and headphones will be worn. Since these headphones are reusable, they will be disinfected before and after each use.
  Interventions: Other: The virtual reality
- The control group (Experimental): No intervention will perform on the control group before the peripheral intravenous catheterization procedure, and the standard peripheral intravenous catheterization procedure will perform.
  Interventions: Other: The virtual reality; Other: The guided imagery

INTERVENTIONS:
Other: The virtual reality — During the PIK application, 3D visual and audio videos of the beach will be played with an Oculus Go brand virtual reality (VR) headset until the procedure is completed. The video that starts at the beginning of the procedure is planned to last approximately 2-3 minutes during the application. During this time, patients will be asked to close their eyes and take a comfortable position. The VR headset will be disinfected after each application and used on the other patient.
  Arms: The control group; The guided imagery group
Other: The guided imagery — Patients in this group will be played an audio clip that helps them imagine walking on a beach and gives instructions during the walk until the procedure is completed, using an MP3 player and headphones. The audio clip aims to activate the imagination of patients by allowing them to use their senses. For example, the temperature of the sun (feeling), the texture of the sand (touching), the color of the sea (seeing), the sound of the waves (hearing), and the smell of the sea (smell) are some examples of this. The audio clip will be voiced by a professional voice artist with good diction. It is planned that the audio clip will be played for approximately 2-3 minutes during the application. During this time, patients will be allowed to close their eyes and take a comfortable position. The headphones of the MP3 player will be disinfected after each application and used on the other patient.
  Arms: The control group; The virtual reality group

SUMMARY:
Aim: The aim of the present study was to examine the effect of virtual reality and guided imagery to reduce pain during peripheral intravenous catheterization procedures in adults.Methods: The study will include 90 adults who were randomly selected between February and March 2025. One application group (n=30) will receive a virtual reality glasses application; the other application group (n=30) will receive a guided imagery application. The applications to the site of the peripheral intravenous catheterization will last two minutes. The control group (n=30) will receive the standard peripheral intravenous catheterization application procedure. The groups' level of pain during catheterization will be assessed using a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Being in accordance with time and place
* Being in no sensory problems
* Being aged between 18 and 65 years
* Being able to evaluate the visual analog scale correctly
* Participating voluntarily in the research.

Exclusion Criteria:

* Not participating voluntarily in the research
* Not fitting the inclusion criteria of the research
* Having a vision or hearing problem
* Having any illness which could affect pain perception, such as sensorymotor disorder, diabetes, peripheral vascular diseases or peripheral neuropathy
* Having phlebitis, scar tissue, dermatitis, an incision or findings of infection at the place where the intervention was to be performed
* Having taken an analgesic (within the previous six hours) or an anesthetic agent before the peripheral intravenous catheterization procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
procedure duration in sec | during the intervention/procedure
  In the stages of the peripheral intravenous catheterization intervention of individuals in the application and control groups, a chronometer will start immediately after an automatic tourniquet is attached to the patient's arm. After catheterization was completed successfully, the chronometer was stopped, and the procedure duration was recorded in the form of seconds on the data collection form.
pain intensity in mm | during the intervention/procedure
  A 10-cm vertical VAS was used to evaluate the severity of pain felt by the individuals during the procedure. The lowest score that can be obtained from the scale is 0 and the highest score is 10 cm (100 mm). Pain severity was evaluated in millimeters
procedure satisfaction in mm | during the intervention/procedure
  A scale between 1 and 10 will be used to evaluate the patients' satisfaction levels with the procedure. "1" on this scale indicates the least satisfaction level, and "10" indicates the highest satisfaction level. Patients will be asked to mark their level.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Cigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided